CLINICAL TRIAL: NCT03274661
Title: Evaluating Immune Checkpoint Inhibition In Solid Tumor Patients With Homologous Recombination Repair Deficiency
Brief Title: Pembrolizumab Activity in Patients With Homologous Recombination Competent and Deficient Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baptist Health South Florida (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Miami Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-3475-663
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Results first posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-09

CONDITIONS: Solid Tumor, Adult
Keywords: solid tumor, Pembrolizumab,
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Eligible participants will receive pembrolizumab intravenously at a dose of 200 mg every 3 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab 200 mg Q3W (Experimental): Pembrolizumab 200 mg Intravenous Infusion every 3 weeks administered on Day 1 of each 3 week cycle
  Interventions: Drug: Pembrolizumab 200 mg Q3W

INTERVENTIONS:
Drug: Pembrolizumab 200 mg Q3W — Pembrolizumab 200 mg Intravenous Infusion every 3 weeks administered on Day 1 of each 3 week cycle
  Other Names: Pembrolizumab 200 mg

SUMMARY:
Phase II trial in which patients with metastatic solid tumors experiencing progression after first line standard chemotherapy or for which there is no standard chemotherapy, and for which pembrolizumab does not have an FDA or compendia listing approved indication, will receive pembrolizumab intravenously at a dose of 200 mg every 3 weeks.

DETAILED DESCRIPTION:
Patients with metastatic or recurrent solid malignancy who have progressed on first line standard of care treatment or for which defined standard of care does not exist or is not readily available are eligible to participate on this trial. Patients for which pembrolizumab has an FDA approved indication and for whom pembrolizumab is covered by their insurance should receive standard commercial pembrolizumab and will not be eligible for this trial.

The primary objective of this trial is to evaluate the Immune-Related Objective Response Rate (IR-ORR) achieved with pembrolizumab in patients with Fanconi Anemia Repair Pathway functionally competent and functionally deficient tumors.

Trial treatment should be administered on Day 1 of each cycle after all procedures/assessments have been completed. Trial treatment may be administered up to 3 days before or after the scheduled Day 1 of each cycle due to administrative reasons.

All trial treatments will be administered on an outpatient basis.

Pembrolizumab 200 mg will be administered as a 30 minute IV infusion every 3 weeks. Target infusion timing is 30 minutes.

Expansion Cohort:

Ten (10) additional subjects with the diagnosis of metastatic or recurrent endometrial carcinoma will be enrolled in the trial at the conclusion of regular enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Have measurable disease based on RECIST 1.1.
* Be willing to provide consent for retrieval of archival tumor material tissue from a previously obtained core or excisional biopsy of a tumor lesion.
* Have a tumor presentation at screening for which pembrolizumab does not have an FDA approved indication for commercial use.
* Have a performance status of 0, 1 or 2 on the ECOG Performance Scale.
* Demonstrate adequate organ function
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication.

Expansion cohort - additional criteria

1. Diagnosis of Endometrial Carcinoma or Sarcoma which is metastatic and has failed standard treatment or is recurrent, or for which standard chemotherapy is contraindicated or refused by patient.
2. Sufficient tissue is available for correlative studies
3. MSI studies have been performed, either by immunohistochemistry or next generation sequencing and results show that patient is MS low or stable.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy, or used an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has a known history of active Bacillus Tuberculosis
* Hypersensitivity to pembrolizumab or any of its excipients.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).
* Has immunohistochemically proven mismatch repair deficient cancer
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Evidence of interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2022-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Diaz, MD, Principal Investigator — Miami Cancer Institute at Baptist Health, Inc.
Locations (1):
- Miami Cancer Institute at Baptist Health, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Villalona-Calero MA, Diaz JP, Duan W, Diaz Z, Schroeder ED, Aparo S, Gatcliffe T, Albrecht F, Venkatappa S, Guardiola V, Garrido S, Rubens M, DeZarraga F, Vuong H. Pembrolizumab activity in patients with Fanconi anemia repair pathway competent and deficient tumors. Biomark Res. 2022 Jun 3;10(1):39. doi: 10.1186/s40364-022-00386-0. PMID 35658948
- See also: MCI - Website — http://baptisthealth.net/cancer-care/home

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab 200 mg Q3W
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab 200 mg Q3W
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 45
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Immune-related Objective Response Rate
Description: Immune-related Response Criteria (irRC) will be utilized for assessment of response to therapy, defined as the percent of participants who achieved complete or partial response. Per irRC, for target lesions assessed by CT or MRI: Complete Response (CR), Disappearance of all lesions in two consecutive observations not less than 4 weeks apart; Partial Response (PR), ≥50% decrease in tumor burden compared with baseline in two observations at least 4 weeks apart.
Time Frame: 20 weeks
Population: Two participants were excluded from analysis: one was deemed not response-evaluable after a further review of baseline CT images demonstrated not clearly measurable disease; another deteriorated rapidly due to tumor progression within a week of the first dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg Q3W
Number analyzed (Participants) | 50
Participants | 9

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Immune-related Response Criteria (irRC) will be utilized for assessment of response to therapy. PFS will be defined as the time from treatment start to time of disease progression or death, whichever comes first. Per irRC, for target lesions assessed by CT or MRI: Progressive Disease (PD), at least 25% increase in tumor burden compared with nadir (at any single time point) in two consecutive observations at least 4 weeks apart.
Time Frame: 20 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Pembrolizumab 200 mg Q3W
Number analyzed (Participants) | 50
months | 2.9 [2.3 to 5.9]

3. Secondary Outcome: Overall Response
Description: Immune-related Response Criteria (irRC) will be utilized for assessment of response to therapy, defined as the duration of time from start of treatment to end of study or death, whichever comes first. Per irRC, for target lesions assessed by CT or MRI:Complete Response (CR) is the disappearance of all lesions in two consecutive observations not less than 4 weeks apart; Partial Response (PR) is a ≥50% decrease in tumor burden compared with baseline in two observations at least 4 weeks apart; and Progressive Disease (PD) is at least 25% increase in tumor burden compared with nadir (at any single time point) in two consecutive observations at least 4 weeks apart. Everything else is considered Stable Disease (SD).
Time Frame: 3 years
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Pembrolizumab 200 mg Q3W
Number analyzed (Participants) | 50
months | 10.9 [5.2 to 21.0]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Pembrolizumab 200 mg Q3W
All-Cause Mortality (participants affected / at risk) | 38/52
Serious Adverse Events (participants affected / at risk) | 19/52
Other Adverse Events (participants affected / at risk) | 30/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg Q3W (N=52)
Abdominal pain (Gastrointestinal disorders) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
Ascites (General disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Stroke (Vascular disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Obstruction - gastric (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Fall (General disorders) | 1 (1)
Urinary retention - Hydronephrosis (Renal and urinary disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Female genital tract fistula - rectovaginal fistula (Reproductive system and breast disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Urinary retention - Urinary tract infection (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Hypercalcemia (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg Q3W (N=52)
Fatigue (General disorders) | 13 (16)
Nausea (Gastrointestinal disorders) | 7 (8)
Constipation (Gastrointestinal disorders) | 8 (8)
Diarrhea (Gastrointestinal disorders) | 3 (6)
Elevated creatinine (Renal and urinary disorders) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Anorexia (Gastrointestinal disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Back pain (General disorders) | 3 (4)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4)
Bloating (Gastrointestinal disorders) | 3 (3)
Elevated lactate dehydrogenase (General disorders) | 3 (3)
Edema (leg) (Cardiac disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Insomnia (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/61/NCT03274661/Prot_SAP_000.pdf